CLINICAL TRIAL: NCT01527825
Title: Immunogenicity and Safety of Different Dosing Schedules of Trivalent Influenza Vaccine in HIV-infected Pregnant Women: a Randomized Controlled Trial
Brief Title: Immunogenicity and Safety of Different Dosing Schedules of Trivalent Influenza Vaccine in HIV-infected Pregnant Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Witwatersrand, South Africa (Other)
Responsible Party: Principal Investigator, Michelle Groome, Senior medical officer, University of Witwatersrand, South Africa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MatfluHIVpos_3dosingschedule
Record Dates: First submitted 2011-12-14; First posted 2012-02-07 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; vaxigrip; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Single dose (Active Comparator): Trivalent Influenza Vaccine (seasonal)
  Interventions: Biological: Trivalent influenza vaccine (seasonal); Biological: Normal saline
- Double dose TIV (Experimental): Trivalent Influenza vaccine (seasonal) Two doses will be administered at enrolment
  Interventions: Biological: Trivalent influenza vaccine (seasonal); Biological: Normal saline
- Two dose TIV (Experimental): Trivalent Influenza vaccine (seasonal) Participants will receive two doses of TIV, one month apart
  Interventions: Biological: Trivalent influenza vaccine (seasonal); Biological: Normal saline

INTERVENTIONS:
Biological: Trivalent influenza vaccine (seasonal) — Single 0.5ml dose of Southern hemisphere 2012 TIV, formulation containing:
  * An A/California/7/2009 (H1N1)pdm-like virus
  * An A/Perth/16/2009 (H3N2)-like virus*
  * A B/Brisbane/60/2008-like virus * A/Wisconsin/15/2009 and A/Victoria/210/2009 are A/Perth/16/2009-like viruses for use in the 2012 Southern Hemisphere winter. This vaccine is the same as the vaccine used for the 2011 Southern hemisphere influenza season.
  Other Names: Vaxigrip
Biological: Normal saline — 0.5ml normal saline will be used as 'placebo' vaccine to maintain blinding
  Other Names: NaCl

SUMMARY:
The overall aim of this project is to evaluate the safety and immunogenicity of 3 different dosing options of trivalent influenza vaccine (TIV) vaccination of HIV-infected pregnant women: single dose, double dose (at same time point) and two-doses (1 month apart).

DETAILED DESCRIPTION:
Determining the contribution of influenza to early childhood morbidity and mortality in sub-Saharan Africa and the potential to prevent influenza disease through vaccination may contribute to reducing childhood deaths; since influenza illness is a vaccine preventable disease for which vaccines are developed, licensed and available at reasonable cost. Unfortunately, infants at highest risk for serious disease are those under 6 months of age, for whom trivalent inactivated influenza vaccine (TIV) is poorly immunogenic and not licensed. As pregnant women also have an increased risk of serious illness (3.3-5.5 fold for hospitalization for influenza-associated acute cardio-respiratory illness) from influenza infection, one strategy to prevent the complications of influenza in pregnant women and young infants is through maternal TIV immunization, which is recommended by the WHO. This could result in direct protection of the women and protection of the young infant consequent to transplacental transfer of TIV induced antibody.

Barriers to administration of vaccines during pregnancy including lack of information on effectiveness and concerns about safety probably explain the virtual non-existent use of TIV in pregnant women from low-middle income countries, including South Africa. Although there was a national campaign for influenza vaccination of pregnant women in South Africa during 2010 due to the concern of continued circulation of H1N1-2009pdm influenza virus, the uptake of vaccine remains poor. TIV immunization of pregnant women is still not provided as standard of care to pregnant women attending antenatal-clinics in South Africa, in part because of absence of any data from any African setting with regard to its risk-benefit ratio.

The immunogenicity and efficacy of TIV in HIV-infected adults was only recently documented in an African setting. This placebo-controlled, community-based randomized, placebo controlled trial, conducted at Themba Lethu HIV clinic, Helen Joseph hospital, reported that TIV was associated with a 75% reduction in influenza-confirmed illness. The results of the study also confirmed the safety of TIV among African HIV-infected adults. The study, however, only included 7 women who were pregnant. In addition to no differences in solicited adverse event rates, there was also no difference in either cluster of differentiation 4 (CD4+) cell count changes or HIV viral control in those on antiretroviral treatment between TIV vaccinees compared to placebo recipients. This allayed previous concerns regarding the potential negative effect of TIV which centered around the observed transient increase in HIV-1 viral load, even in HIV infected individuals on ART and who were virologically suppressed (viral load <400 copies/ml). Decreases in CD4+ lymphocyte counts have also been observed in HIV-infected individuals post TIV vaccination. These changes, however, even in past studies were infrequent (4-18%) and resolved at later time-points and were considered to be clinically non-significant.

Only recently has data become available from another low-income country (Bangladesh) in which the benefit of maternal TIV vaccination was demonstrated by a 63% (95% confidence interval (CI) 5 to 85) reduction in laboratory-confirmed influenza illness in infants under 24 weeks of age in children born to mothers vaccinated with TIV and a 36% reduction in clinical illness in vaccinated mothers. There has, however, not been any study on the effectiveness of maternal immunization with TIV on influenza- associated morbidity and mortality either in the mothers or infants in African settings.

Much of influenza virus associated morbidity and mortality may be due to the synergistic lethality of influenza with bacterial pathogens leading to pneumonia as well as other viral co-infections. Superimposed bacterial infections, especially Streptococcus pneumoniae and in patients treated with antibiotics, Staphylococcus aureus, contribute to a large proportion (28-65%) of pneumonia deaths associated with influenza illness during pandemics. Unpublished data from the Bangladeshi study show that infants of mothers who received TIV (with pneumococcal conjugate vaccine, 7 valent (PCV7) given to infants) were better protected from acquisition of pneumococcal carriage during influenza season than infants of TIV-unimmunized mothers. No data in the African setting are available to support or refute this observation from Bangladesh. As introduction of pneumococcal conjugate vaccines (PCV) in low-income countries is a priority of the Global Alliance for Vaccines and Immunization (GAVI), with 7 African countries already approved, and many others to follow, to introduce PCV within the next five years.

Despite the encouraging results on maternal immunization from Bangladesh, and the preliminary data supporting that TIV is efficacious mainly in HIV-infected non-pregnant adults, further data are needed to advocate for routine use of TIV during pregnancy in settings with a high prevalence of HIV. Reasons for this include that the impact of maternal HIV on the kinetics of TIV induced transplacental antibody transfer cannot be derived from available data. This is important as the primary focus of this proposal, and major potential public health benefit of maternal TIV vaccination, is targeted at protection of young infants. HIV infection is known to decrease placental integrity and lower antibody levels in the fetus and newborn. Furthermore, maternal hypergamma-globulinemia that is characteristic of HIV-infection may be associated with decreased neonatal antibody levels. This paradox is explained by the limited number of placental antibody receptors, resulting in immunoglobulin G (IgG) antibodies competing for available receptors and thereby decreasing vaccine-specific antibody transport. Preterm birth increases with HIV, chronic maternal disease or malnutrition. Transfer of maternal antibody which is gestational age dependant, may be more affected by maternal immunization in sub-Saharan Africa where these conditions are common.

In 2011, two Maternal influenza vaccination trials are being conducted in pregnant women from the Soweto community, one in HIV-infected women, and the other in HIV-uninfected women. In both these trials (HREC reference number 101106 and 101107) the immunogenicity of a single dose of TIV administered between 20 and 36 weeks of gestation was investigated.

HIV-uninfected women showed a good response one month post vaccination with 85.3%, 92.7% and 98.5% of women having seroprotective levels of antibodies to the vaccine strains, H3N2, H1N1 and B respectively, however, HIV-infected women showed an inferior response to vaccination. The CD4+ cell count at baseline (prior to vaccination) affected the immunological response mounted by HIV-infected women: 12.5%, 12.5% and 62.5% of women with CD4+ cell count <200, and 50%, 66.7% and 77.8% of women with CD4+ count ≥500 had seroprotective levels to vaccine strains, H3N2, H1N1 and B respectively, one month post receipt of single-dose TIV.

The overall aim of this project is to evaluate the safety and immunogenicity of 3 different dosing options of TIV vaccination of HIV-infected pregnant women: single dose, double dose (at same time point) and two-doses (1 month apart)

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women age under 18 years to under 39 years.
* Gestational age greater or equal 12 weeks to under 36 weeks documented by the approximate date of the last menstrual period and corroborated by physical/ sonar examination.
* Documented to be HIV-infected on two assays prior to study-enrolment.
* Able to understand and comply with planned study procedures.
* Provides written informed consent prior to initiation of study.

Exclusion Criteria:

* Features of WHO clinical category 3 or 4 of AIDS at the time of enrolment.
* Receipt of TIV, other than through the study, during the current influenza season documented by medical history or record.
* Receipt of any live licensed vaccine 28 days or less or inactivated licensed vaccine (EXCEPT tetanus toxoid) 14 days or less prior to study-vaccine.
* Receipt of a non-licensed agent (vaccine, drug, biologic, device, blood product, or medication) 28 days or less prior to vaccination in this study, or expects to receive another non-licensed agent before delivery unless study approval is obtained.
* Any significant (in the opinion of the site investigator) acute illness and/or oral temperature greater than or equal to 38 degrees Celcius ≤ 24 hours prior to study entry.
* Use of anti-cancer systemic chemotherapy or radiation therapy ≤ 48 weeks of study enrollment, or has immunosuppression as a result of an underlying illness or treatment.
* Long term use of glucocorticoids, including oral or parenteral prednisone ≥ 20 mg/day or equivalent for more than 2 consecutive weeks (or 2 weeks total) ≤ 12 weeks of study entry, or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) ≤ 12 weeks before study entry (nasal and topical steroids are allowed).
* Receipt of corticosteroids for preterm labor ≤ 14 days before study entry.
* Receipt of immunoglobulin or other blood products (with exception of Rho D immune globulin) ≤ 12 weeks prior to enrollment in this study or is scheduled to receive immunoglobulin or other blood products (with the exception of Rho D immune globulin) during pregnancy or for the first 24 weeks after delivery.
* Receipt of interleucin 2 (IL2), interferon (IFN), GMCSF or other immune mediators ≤ 12 weeks before enrollment.
* Uncontrolled major psychiatric disorder.
* History of a severe adverse reaction to previous TIV.
* Any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
* Pregnancy complications (in the current pregnancy) such as pre-term labor, hypertension (BP >140/90 in the presence of proteinuria or BP >150/100, with or without proteinuria or currently on antihypertensive medication) and pre-eclampsia.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 800 (Actual)
Dates: Start 2012-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Number of participants who mount an adequate immune response one month post vaccination to a double dose compared to single dose of TIV | One month (28-35 days) post vaccination
  Determine the sero-response rate to each of the vaccine viral strains, defined as post vaccination hemagglutination inhibition (HAI) levels of ≥1:40 AND ≥4 fold increase over baseline HAI levels, in HIV-infected pregnant women receiving a double strength TIV dose compared to mothers receiving a single dose of TIV one-month after completion of the dosing schedule.
Number of participants who mount an adequate immune response one month post completing vaccination to two-dose TIV administered 1 month apart, compared to single dose TIV | One month (28-35 days) post vaccination
  Determine the sero-response rate to each of the vaccine viral strains, defined as post vaccination HAI levels of ≥1:40 AND ≥4 fold increase over baseline HAI levels, in HIV-infected pregnant women receiving two-doses of TIV spaced 21-35 days apart compared to women receiving a single dose of TIV one-month after completion of the dosing schedule.
Number of participants in each treatment arm who have local and/ or systemic reactions post vaccination with TIV | One week post vaccination
  Evaluate the safety of the three dosing schedules of TIV in HIV-infected pregnant women vaccinated between 12-36 weeks of gestational age.

SECONDARY OUTCOMES:
Number of infants born to mothers who received double- or two doses of TIV who are seroprotected against influenza compared to infants born to mothers in single dose arm. | Within first week of life (0-7 days)
  Compare the proportion of newborns born to HIV-infected mothers in the double dose and two-dose arms with HAI antibody titers of ≥1:40 to each of the three TIV strains to newborns of HIV-infected and HIV-uninfected women (enrolled in separate parallel cohort) who received single dose of TIV.
Number of infants with protective maternal antibody levels against TIV at birth and at 8, 16 and 24 weeks of age | Birth to 24 weeks post delivery
  Determine the kinetics of transplacental transfer of maternal Hemagglutinin (HA) antibodies and persistence thereof until 24 weeks post-partum in the infants.
Number of infants born to women in double- and two dose TIV arms, compared to single TIV dose arm who are protected against laboratory confirmed influenza | Birth to 24 weeks
  Compare the relative efficacy of a double-strength or two-dose dose TIV schedule compared to a single dose TIV schedule in pregnant HIV-infected women in protecting against laboratory-confirmed influenza illness in their infants up to 24 weeks of chronological age.
Number of infants born to women in double- and two- dose TIV arms compared to single dose arm who are protected against clinical influenza like illness | Birth to 24 weeks post delivery
  Compare the relative efficacy of a double-strength or two-dose dose TIV schedule compared to a single dose TIV schedule in pregnant HIV-infected women in protecting against protocol defined clinical influenza like illness (ILI) in their infants up to 24 weeks of chronological age.
Number of women protected against laboratory confirmed influenza in each treatment arm | From date of vaccination (12 to 36 weeks gestational age [GA]) until infant is 24 weeks old. Anticipated mean GA at randomisation is 20 weeks, and at delivery is 39 weeks, so average follow up period is 43 weeks, however it could be as long as a year.
  Compare the relative efficacy of a double-strength or two-dose dose TIV schedule compared to a single dose TIV schedule in pregnant HIV-infected women in protecting against laboratory-confirmed influenza illness in maternal participants up to 24 weeks post partum.
Number of women protected against clinical influenza like illness in each treatment arm | From date of vaccination (12 to 36 weeks gestational age [GA]) until infant is 24 weeks old. Anticipated mean GA at randomisation is 20 weeks, and at delivery is 39 weeks, so average follow up period is 43 weeks, however it could be as long as a year.
  Compare the relative efficacy of a double-strength or two-dose dose TIV schedule compared to a single dose TIV schedule in pregnant HIV-infected women in protecting against protocol defined clinical ILI in maternal participants up to 24 weeks post partum.
Number of women who mount immune responses (seroconversion /seroprotection)in each treatment arm | From date of vaccination (12 to 36 weeks gestational age [GA]) until infant is 24 weeks old. Anticipated mean GA at randomisation is 20 weeks, and at delivery is 39 weeks, so average follow up period is 43 weeks, however it could be as long as a year.
  Define and compare cell mediated immune responses to different dosing options of TIV in HIV-infected pregnant women.
Number of women who have changes to CD4+ and/ or viral load results post vaccination in each treatment arm | From date of vaccination (12 to 36 weeks gestational age [GA]) until infant is born. Anticipated mean GA at randomisation is 20 weeks, and at delivery is 39 weeks, so average follow up period is 19 weeks, however it could be as long as 30 weeks.
  Evaluate the effect of TIV (single, double and two doses) on CD4+ cell count and HIV-viral load changes comparing baseline levels to levels at delivery.
Number of participants in each treatment arm who suffer adverse pregnancy outcomes (maternal or foetal) after TIV-vaccination | From date of vaccination (12 to 36 weeks gestational age [GA]) until infant is born. Anticipated mean GA at randomisation is 20 weeks, and at delivery is 39 weeks, so average follow up period is 19 weeks, however it could be as long as 30 weeks.
  Describe safety outcome measures (maternal and foetal) of TIV-vaccination of HIV-infected pregnant women

CONTACTS AND LOCATIONS:
Overall Officials: Shabir A Madhi, MD PhD, Study Chair — University of Witwatersrand, South Africa
Locations (1):
- Respiratory and Meningeal Pathogens research unit, Soweto, Johannesburg, Gauteng, South Africa

REFERENCES:
- [Derived] Nunes MC, Cutland CL, Moultrie A, Jones S, Ortiz JR, Neuzil KM, Klugman KP, Simoes EAF, Weinberg A, Madhi SA; Maternal Flu Trial Team. Immunogenicity and safety of different dosing schedules of trivalent inactivated influenza vaccine in pregnant women with HIV: a randomised controlled trial. Lancet HIV. 2020 Feb;7(2):e91-e103. doi: 10.1016/S2352-3018(19)30322-4. Epub 2020 Jan 3. PMID 31911146